CLINICAL TRIAL: NCT07070089
Title: BosSTENT ImpLant to trEat debilitatiNg Pulse-synchronous Tinnitus
Brief Title: BosSTENT Implantation to Treat Pulse-Synchronous Tinnitus
Acronym: B-SILENT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sonorous NV, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-001SON
Record Dates: First submitted 2025-07-03; First posted 2025-07-17 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Pulsatile Tinnitus; Venous Sinus Stenosis
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- BosSTENT (Experimental)
  Interventions: Device: BosSTENT implantation

INTERVENTIONS:
Device: BosSTENT implantation — BosSTENT implantation in the transverse venous sinus

SUMMARY:
This study is evaluating the safety and clinical performance of the BosSTENT, a new stent designed specifically for treating pulse-synchronous tinnitus due to venous sinus stenosis. The study will evaluate the long-term safety of the BosSTENT as well as its impact on the severity of pulse-synchronous tinnitus.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 - 80 years old
2. Able to provide informed consent to participate in the study
3. Severe or catastrophic PST (THI grade ≥ 4; THI score ≥ 58) that responds to jugular vein compression.
4. Cerebral venous sinus stenosis with the following characteristics:

   1. Transverse cerebral venous sinus
   2. >50% stenosis by computed tomography venogram (CTV), magnetic resonance venogram (MRV), or catheter cerebral angiography
   3. Vessel diameter amenable to sizing according to Table 1 below without the need to undersize
5. Attempted PST amelioration with at least one non-invasive therapy (i.e., refractory to non-invasive therapy)
6. Willing to comply with protocol requirements and return to the treatment center for all required clinical evaluations and follow-up
7. Life expectancy >12 months

Exclusion Criteria:

1. Dural cerebral venous sinus stenosis secondary to an underlying condition (e.g. brain tumor) that may be treated by alternative established therapies (e.g., surgery, embolization)
2. Previously implanted stent in the target vessel
3. Contraindication to anticoagulant and/or antiplatelet therapy or thrombolytic drugs
4. Target vessel size that does not fall within the indicated range per Table 1 of the IFU
5. History of severe allergy to contrast/contrast media or nickel
6. Non-pulse-synchronous tinnitus
7. Current diagnosis of papilledema
8. Dural arteriovenous fistula or arteriovenous malformation
9. History of untreated atrial fibrillation, untreated/uncontrollable hypertension, or other stroke factors
10. History of deep vein thrombosis or pulmonary embolism
11. History of heart failure, dilated cardiomyopathy, or congenital heart conditions
12. Arterial stenosis, dissection, or aneurysm
13. PST due to causes not related to cerebral venous sinus stenosis
14. Evidence of an active systemic infection
15. Venous sinus thrombosis, jugular compression, venous aberrant or tortuous anatomy that would prevent the safe delivery and deployment of the BosSTENT to the target treatment zone.
16. Cerebral venous sinus diverticulum that, in the Investigator's opinion, requires treatment other than stenting (e.g., coiling)
17. Otologic disorders that may confound PST assessments, including, but not limited to misophonia or hyperacusis
18. Hypercoagulable state or hemorrhagic or coagulation deficiency refractory to medical therapy
19. Suffered a stroke within the past 6 months
20. Platelet count <100x109/L (100,000/µL)
21. Participation in another investigational protocol
22. Immuno-compromised
23. Pregnant or nursing women (females of childbearing potential who are less than 45 years old must have a pregnancy test and provide written proof that they are not pregnant prior to inclusion)
24. Other clinical conditions, that in the opinion of the Investigator significantly compromise the ability to perform a safe and/or effective procedure
25. Incapacitated, mentally compromised or otherwise incapable of understanding and/or providing informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major adverse events (MAE) | 3 months
  MAEs are defined as symptomatic, serious, procedure- or device-related post-procedure complications: major stroke, neurological death, in-stent thrombosis, target vessel restenosis, stent-adjacent stenosis, or stent migration
Improvement of pulse-synchronous tinnitus measured by a decrease of at least 2 grades or 40 points on the Tinnitus Handicap Inventory (THI) | 30 days
  THI ranges from 0-100 points with zero indicating no handicap due to tinnitus and increasing scores indicating progressively worse handicap due to tinnitus. Grades range from 1-5 going from Slight (0-16 points), to Mild (18-36 points), Moderate (38-56 points), Severe (58-76 points) and finally Catastrophic (78-100 points)

IPD SHARING:
Plan to Share IPD: No
This study is intended to determine incidences of major adverse events and pulse-synchronous tinnitus improvement. While specific events may be summarized in study reports or publications, IPD are not anticipated to be shared.